CLINICAL TRIAL: NCT05429359
Title: cArdiopulmonary exerCise Test Assessing Multiple biOmarkers and Hormones iN Type 1 diabetEs Under Different Circumstances (ACT-ONE)
Brief Title: cArdiopulmonary exerCise Test Assessing Multiple biOmarkers and Hormones iN Type 1 diabetEs Under Different Circumstances
Acronym: ACT-ONE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Universiteit Antwerpen (Other); York University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ACT-ONE
Record Dates: First submitted 2022-06-17; First posted 2022-06-23 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-06

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: exercise; biomarker; glucose; lactate; ketones; continuous glucose monitoring; hormones
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity; Ketosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CSII users (Active Comparator): Patients using Continuous Subcutaneous Insulin Infusion (only hybrid closed loop pumps)
  Interventions: Other: CPET: CardioPulmonary Exercise Test for CSII users; Other: AEX1: Aerobic Exercise Test 1 for CSII users; Other: AEX2: Aerobic Exercise Test 2 for CSII users
- MDI users (Active Comparator): Patients using Multiple Daily Injections (only Tresiba and Toujeo as basal insulin)
  Interventions: Other: CPET: CardioPulmonary Exercise Test for MDI users; Other: AEX1: Aerobic Exercise Test 1 for MDI users; Other: AEX2: Aerobic Exercise Test 2 for MDI users

INTERVENTIONS:
Other: CPET: CardioPulmonary Exercise Test for CSII users — * Baseline
  * VO2peak measurement
  * Breakfast
  * 100% bolus insulin
  * CSII users: 100% basal
  Arms: CSII users
Other: AEX1: Aerobic Exercise Test 1 for CSII users — * 90min
  * 40-45% VO2peak
  * Breakfast
  * 50% bolus insulin
  * CSII users: -2h target 150 mg/dL
  Arms: CSII users
Other: AEX2: Aerobic Exercise Test 2 for CSII users — * 90min
  * 40-45% VO2peak
  * Breakfast
  * 50% bolus insulin
  * CSII users: -1h target 150 mg/dL
  Arms: CSII users
Other: CPET: CardioPulmonary Exercise Test for MDI users — * Baseline
  * VO2peak measurement
  * Breakfast
  * 100% bolus insulin
  * MDI users: 100% basal
  Arms: MDI users
Other: AEX1: Aerobic Exercise Test 1 for MDI users — * 90min
  * 40-45% VO2peak
  * Breakfast
  * 50% bolus insulin
  * MDI users: 50% basal
  Arms: MDI users
Other: AEX2: Aerobic Exercise Test 2 for MDI users — * 90min
  * 40-45% VO2peak
  * Breakfast
  * 50% bolus insulin
  * MDI users: 80% basal
  Arms: MDI users

SUMMARY:
Collection of venous blood samples in 50 persons with type 1 diabetes to evaluate the behavior of different biomarkers (glucose, lactate, beta-hydroxybutyrate), and hormones (cortisol, growth hormone) during and after one morning CardioPulmonary Exercise Test and 2 aerobic (90 minutes at 40-45% of VO2 max) exercise tests under different circumstances (see Protocol).

DETAILED DESCRIPTION:
This study is an extension of the Action-1 pilot study. This study is an extension of the Action-1 pilot study. The aim is to collect samples of multiple biomarkers (circulating glucose, ketones and lactate levels) and hormones (cortisol and growth hormone) during and following an anaerobic and two aerobic exercise in patients with T1D, under more and well-defined circumstances (bolus insulin reduction in combination with major vs. minor basal insulin reduction) to aim for safer glucose levels during and after exercise (~90-180 mg/dL or ~5-10 mmol/L) and avoid extreme glucose excursions to hypo (< 70 mg/dL or <3.9 mmol/L) or hyperglycemia (>180 mg/dL or >10 mmol/L). Based on these data, we aim to formulate exercise guidelines to better help prevent hypoglycemia during and after exercise. Overall, our goal is to help maintain target glycemic values during and after exercise, as evidenced by >70% time in range (70-180mg/dL) while using Continuous Glucose Monitoring (CGM).

Primary endpoint:

• CGM outcomes during and after morning exercise, determined as:

* Time in range (TIR) 70-180mg/dL
* Time below range (TBR) Level 2, <54 mg/dL
* Time below range (TBR) Level 1 and 2, <70 mg/dL
* Time above range (TAR) Level 1 and 2, >180 mg/dL
* Time above range (TAR) Level 2, >250 mg/dL

Secondary endpoints:

* Evaluate values and trends of glucose, lactate and beta-hydroxybutyrate before, during and after morning exercise in venous blood.
* Evaluate trends of cortisol and growth hormone before, during and after exercise in relationship to possible hypoglycemic (<70mg/dL glucose) and hyperglycemic events (>180mg/dL).

One CardioPulmonary Exercise Test (CPET, symptom limited maximal exercise test) and two Aerobic Exercise Tests at 40-45% VO2max (AEX), with venous blood samples (catheter), heart rate monitoring during the exercise and follow-up to 6h after the exercise.

(The individual VO2max, using a CardioPulmonary Exercise Test, can be determined during the first "Symptom Limited Maximal" Exercise Test. This to assess the VT1 (V-slope relation VCO2 and VO2; Eq02), VT2 (Relation VE and VCO2; EqCO2) and VO2 peak.)

Before exercise Test 1, the CPET, the study participants will receive 7 questions on the physical activity over the last 7 days (IPAQ questionnaire).

The 3 Exercise Tests will be carried out with 2-4 weeks intervals:

* The day before an exercise test and right before, no exercise (only ADL) is allowed (patients should not come to the study center by bike)
* The night before the exercise test, no hypoglycemia must occur, as defined by 15 consecutive minutes, or more, of an interstitial glucose <70 mg/dL
* Target glucose level in the morning: 90-180 mg/dL
* The morning of the exercise test: patients will receive a standardized breakfast (slices of bread with protein spread (containing ±5-25g of protein in total) of in total 0.5g carbohydrates per kg body weight)
* Breakfast at 30 minutes before the exercise with a bolus at the start of the breakfast (100% bolus for CPET, 50% bolus for AEX)
* Pump settings: basal insulin reduction through temporary target of 150 mg/dL during AEX1 and AEX2 will be adjusted 60-120 minutes prior to the start of the exercise and will last until 60 minutes after the exercise (210-270 min in total)
* Lunch (slices of bread with protein spread (containing ±5-25g of protein in total) of in total 0.5g carbohydrates per kg body weight) will be served after 2h of follow-up with a 75% insulin bolus and a correction bolus, if necessary, of 50% of the patient's usual insulin correction dose for the level of hyperglycemia observed.
* Hyperglycemia (>250mg/dL) before, during and after exercise will be corrected according to the patient's treatment schedule at 50% of the patient's usual correction factor.
* Glucose levels below the target glucose of 90 mg/dL during exercise will be corrected with fast-acting carbohydrates: 15g of oral glucose (sports beverage Aquarius Red Peach (7.4g CHO/100ml)), as repeated every 15 minutes, if necessary, until interstitial and/or whole blood glucose is > 70 mg/dL.

CPET:

* Baseline
* VO2peak measurement
* Breakfast
* 100% bolus insulin
* CSII: 100% basal
* MDI: 100% basal

AEX1:

* 90min
* 40-45% VO2peak
* Breakfast
* 50% bolus insulin
* CSII: -2h target 150 mg/dL
* MDI: 50% basal

AEX2:

* 90min
* 40-45% VO2peak
* Breakfast
* 50% bolus insulin
* CSII: -1h target 150 mg/dL
* MDI: 80% basal

CPET = CardioPulmonary Exercise Test; AEX = Aerobic Exercise Test; CSII = Continuous Subcutaneous Insulin Infusion (only hybrid closed loop pumps); MDI = Multiple Daily Injections (only Tresiba and Toujeo as basal insulin)

ELIGIBILITY:
Inclusion Criteria:

* Duration of type 1 diabetes mellitus >5y
* Subjects willing to sign an informed consent form (ICF)
* Age 18-60y
* Using a continuous glucose monitoring system (preferably Guardian or Dexcom for CSII / Freestyle Libre for MDI)
* For CSII: only hybrid closed loop pumps (HCL)
* For MDI: only Tresiba (degludec) & Toujeo (glargine)
* HbA1c 6-8.0% (blood result up to 3 months old)
* BMI 20-27.5 kg/m2
* The participant should be in the categories 'moderately' to 'highly physically active' according to the IPAQ score
* The Physical Activity Coefficient has not changed (from category1) in the 2 months prior to the first Exercise Test

Exclusion Criteria:

* Being pregnant or having an active pregnancy wish
* Subject not on MDI or CSII
* Musculoskeletal disorder that affects cycling or is a contra-indication for vigorous physical activity
* Cardiorespiratory disease or ECG abnormality that is a contra-indication for vigorous physical activity
* Having an acute illness (e.g. influenza) that interferes with glucose metabolism
* Having a metabolic disorder (different from diabetes) known to have significant interference with glucose metabolism
* Current treatment with drugs known to have significant interference with glucose metabolism, such as systemic corticoids as judged by the investigator
* Presence of concomitant pathology such as heart failure, liver failure, kidney failure (defined as eGFR <45mL/min, blood result up to 12 months old)
* (Severe) food allergies as judged by the investigator

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
CGM outcomes during and after morning exercise | CGM values will be collected up to 8 hours prior to the exercise test and 24 hours after the exercise test
  CGM outcomes, determined as:
  * Time in range (TIR) 70-180mg/dL
  * Time below range (TBR) Level 2, <54 mg/dL
  * Time below range (TBR) Level 1 and 2, <70 mg/dL
  * Time above range (TAR) Level 1 and 2, >180 mg/dL
  * Time above range (TAR) Level 2, >250 mg/dL

SECONDARY OUTCOMES:
Change in glucose concentration in venous blood during and after morning exercise test | Blood sampling was done before the exercise, every 3-10 minutes during the exercise and every 15 minutes during the first hour of recovery and every 30-60 minutes during the rest of the 6-hour follow-up
  Glucose levels in mg/dL during and after CardioPulmonary Exercise Test and 2 morning Aerobic Exercise Tests (90 minutes at 40-45% of VO2 max) (CPET & AEX1-2), measured through EKF
Change in lactate concentration in venous blood during and after morning exercise test | Blood sampling was done before the exercise, every 3-10 minutes during the exercise and every 15 minutes during the first hour of recovery and every 30-60 minutes during the rest of the 6-hour follow-up
  Lactate levels in mM during and after CardioPulmonary Exercise Test and 2 morning Aerobic Exercise Tests (90 minutes at 40-45% of VO2 max) (CPET & AEX1-2), measured through EKF
Change in ketone concentration in venous blood during and after morning exercise test | Blood sampling was done before the exercise, every 3-10 minutes during the exercise and every 15 minutes during the first hour of recovery and every 30-60 minutes during the rest of the 6-hour follow-up
  Ketone (Beta-hydroxybutyrate) levels in mM during and after CardioPulmonary Exercise Test and 2 morning Aerobic Exercise Tests (90 minutes at 40-45% of VO2 max) (CPET & AEX1-2), measured through EKF
Change in cortisol concentration in venous blood during and after morning exercise test | Blood sampling was done before the exercise, every 15-30 minutes during the exercise and every 15-30 minutes during the first hour of recovery and every 60-120 minutes during the rest of the 6-hour follow-up
  Cortisol levels during and after CardioPulmonary Exercise Test and 2 morning Aerobic Exercise Tests (90 minutes at 40-45% of VO2 max) (CPET & AEX1-2), measured through venous blood sampling analysis
Change in growth hormone concentration in venous blood during and after morning exercise test | Blood sampling was done before the exercise, every 15-30 minutes during the exercise and every 15-30 minutes during the first hour of recovery and every 60-120 minutes during the rest of the 6-hour follow-up
  Growth hormone levels during and after CardioPulmonary Exercise Test and 2 morning Aerobic Exercise Tests (90 minutes at 40-45% of VO2 max) (CPET & AEX1-2), measured through venous blood sampling analysis

CONTACTS AND LOCATIONS:
Overall Officials: Christophe De Block, MD, PhD, Principal Investigator — University Hospital, Antwerp

IPD SHARING:
Plan to Share IPD: No